CLINICAL TRIAL: NCT01305668
Title: Effectiveness of Pulmonary Rehabilitation in Chronic Obstructive Pulmonary Disease (COPD) Patients With Emphysema Phenotype
Brief Title: Rehabilitation in Chronic Obstructive Pulmonary Disease (COPD) Patients With Emphysema
Status: Completed | Type: Observational
Sponsor: Villa Pineta Hospital (Other)
Responsible Party: Principal Investigator, Prof. Clini Enrico, Villa Pineta Hospital, Villa Pineta Hospital
Other Study IDs: VP-01-2011
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema
Keywords: COPD; Emphysema phenotype
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Emphysema phenotype
- No-Emphysema phenotype

SUMMARY:
Chronic Obstructive Pulmonary Disease has two heterogeneous conditions (chronic bronchitis and pulmonary emphysema phenotypes) with a different clinical presentation.

The phenotype evaluation in COPD patient (trough clinical, functional and radiographic parameters) could influence final results in pharmacologic and non-pharmacologic management of the disease.

The aim of our study is to investigate whether COPD patients with different disease phenotype (chronic bronchitis versus pulmonary emphysema) have a different response to PR.

ELIGIBILITY:
Inclusion Criteria:

* COPD disease with any functional grade
* Adherence to participate to a pulmonary rehabilitation program

Exclusion Criteria:

* Recent acute exacerbation (4 weeks preceding enrollment)
* Acute severe concomitant cardiovascular diseases
* Concomitant neoplastic diseases
* NO-Adherence to participate to a pulmonary rehabilitation program

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with or without Emphysema phenotype
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance | [Time Frame: Day 1 and 20 ]
  Change in Six minute walked distance (6MWD)

SECONDARY OUTCOMES:
Dyspnoea | [ Time Frame: Day 1 and 20]
  Change in dyspnea grade by MRC
Symptoms on effort | [ Time Frame: Day 1 and 20]
  Change in Dyspnoea and leg fatigue by Borg scale
Perceived Quality of life | [ Time Frame: Day 1 and 20]
  Change in Saint George Respiratory Questionnarie (Italian version)
Global function | [ Time Frame: Day 1 and 20]
  Change in the multidimensional BODE index (validated in COPD population)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico M Clini, MD, Study Director — Villa Pineta Hospital and University of Modena and Reggio Emilia
Locations (5):
- Italy (5):
  - Fondazione Maugeri IRCCS, Lumezzane, Brescia
  - Villa Pineta Hospital, Pavullo nel Frignano, Modena
  - Auxilium Vitae Rehabilitation Center, Volterra, Pisa
  - Ospedale San Raffaele, Velletri, Roma
  - Clinic Center, Naples